CLINICAL TRIAL: NCT06592781
Title: Assessing the Knowledge and the Willingness to Accept Renal Transplantation As a Treatment Option Among CKD Patients ,a Cross-sectional Study
Brief Title: Assessing the Knowledge and the Willingness to Accept Renal Transplantation As a Treatment Option Among CKD Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Andrew Al Amir Asham Shafiq, Assistant Lecturer, Assiut University
Other Study IDs: Kidney transplantation in CKD
Record Dates: First submitted 2024-09-08; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Assessing the Knowledge and the Willingness to Accept Renal Transplantation As a Treatment Option Among CKD Patients, a Cross-sectional Study

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Assessing the knowledge and the willingness to accept renal transplantation as a treatment option among CKD patients, a cross-sectional study

DETAILED DESCRIPTION:
Kidney transplantation in CKD patient

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Patients diagnosed to have CKD stage III- stage V (including patients undergoing regular haemodialysis) regardless the duration of the disease

Exclusion Criteria:

* CKD patients of stage I or II of the disease
* Patients with AKI
* Patients refusing to answer the questionnaire
* Patients who are unable to understand the questionnaire
* Patients underwent kidney transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Age >18 years
  2. Patients diagnosed to have CKD stage III- stage V (including patients undergoing regular haemodialysis) regardless the duration of the disease
Sampling Method: Non-Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 2024-09-10 (Estimated); Primary Completion 2025-09-10 (Estimated); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
Assessment of the knowledge and the willingness of CKD patients to accept kidney transplantation | 18 months
  assessment CKD patients' knowledge and willingness about kidney transplantation

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boima V, Amissah-Arthur MB, Yorke E, Dey D, Fiagbe D, Yawson AE, Nonvignon J, Mate-Kole CC. Determinants of willingness to accept kidney transplantation among chronic kidney disease patients in Ghana. BMC Nephrol. 2021 Apr 13;22(1):129. doi: 10.1186/s12882-021-02335-9. PMID 33849488